CLINICAL TRIAL: NCT00868491
Title: Induction Chemotherapy Followed by Chemoradiation With Cetuximab and Cisplatin for Inoperable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Induction Chemotherapy Followed by Chemoradiation With Cetuximab in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR-62202-717
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; inoperable; induction chemotherapy; concomitant radiochemotherapy; biological agent; efficacy; toxicity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- induction chemotherapy plus chemo-immuno-radiotherapy (Experimental): TPF induction chemotheraopy, radiotehrapy, concomitant cisplatin and cetuximab
  Interventions: Drug: docetaxel, cisplatin, 5-fluorouracil; Radiation: radiotherapy; Drug: cetuximab, cisplatin

INTERVENTIONS:
Drug: docetaxel, cisplatin, 5-fluorouracil — docetaxel 75 mg/m2 I.V. day 1, cisplatin 75 mg/m2 I.V. day 1, 5-fluorouracil 750 mg/m2 I.V. continuous infusion days 1-5 repeated every 21 days for 4 cycles
Radiation: radiotherapy — Three-dimensional conformal radiotherapy planning and delivery (35x2 Gy/day over 7 weeks - weeks 14 - 20 of the study protocol
Drug: cetuximab, cisplatin — * cetuximab 400 mg/m2 I.V. week 13, cetuximab 250 mg/m2 I.V. weeks 14-20
  * cisplatin 30 mg/m2 I.V. weeks 14-20 (concomitantly with radiothrapy)
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to determine the efficacy and toxicity of docetaxel/cisplatin/5-fluorouracil induction chemotherapy (4 cycles) followed by concomitant chemoradiation with cetuximab and weekly cisplatin in patients with inoperable squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
The treatment results with radiotherapy in inoperable squamous cell carcinoma of the head and neck are poor.

In this proposed single-institution non-randomized, one-arm, open label phase II study, the authors will test the efficacy and toxicity of docetaxel/cisplatin/5-fluorouracil induction chemotherapy (4 cycles) followed by concomitant chemoradiation with cetuximab and weekly cisplatin in patients with inoperable squamous cell carcinoma of the head and neck.

Chemotherapy doses will be as follows: docetaxel 75 mg/m2 I.V. day 1, cisplatin 75 mg/m2 I.V. day 1, 5-fluorouracil 750 mg/m2 I.V. continuous infusion days 1-5 repeated every 21 days for 4 cycles followed by cetuximab 400 mg/m2 I.V. week 13, cetuximab 250 mg/m2 I.V. weeks 14-20, cisplatin 30 mg/m2 I.V. weeks 14-20. Three-dimensional conformal radiotherapy planning and delivery (35x2 Gy/day over 7 weeks {weeks 14 - 20}) will be used.

The planned number of patients to be included is 30 and anticipated enrolment period is 12 months.

The primary objective of the study is to determine locoregional control at 2 years post-therapy, whereas secondary objectives are to determine feasibility (toxicity profile) of the proposed regimen, to determine complete response rate after induction ChT as well as 14-16 weeks after the therapy, completion of ChRT to determine disease free survival at 2 years, overall survival at 2 years and late toxicity including thyroid function.

Given the preliminary nature of the study, no stopping rule is prospectively planned outside of observed toxicity, which will be assessed and graded according to Common Terminology Criteria for Adverse Events version 3.0.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma, histologically proven
* Tumour site: oral cavity, oropharynx, hypopharynx or larynx.
* Locally and/or regionally inoperable tumors (UICC TNM stages IVa or IVb) - - without distant metastases (M0-stage)
* Male or female ≥18 years of age
* Expected survival >6 months
* Presence of at least one bidimensionally measurable index lesion
* Effective contraception for both male and female subjects if risk of conception exists
* WHO performance status 0-2
* Laboratory parameters:

hemoglobin ≥100 g/L leukocyte count > 3.5x109/L, absolute neutrophil count ≥ 1.5x109/L platelet count > 100x109/L total bilirubin < 1.25x upper normal limit transaminases (ALT, AST) < 5x upper normal limit creatinine clearance ≥ 55 mls/minute

* Signed written informed consent

Exclusion Criteria:

* Metastatic disease
* Squamous cell carcinoma of the nasopharynx and nasal cavity and paranasal sinuses
* ChT or XRT ineligibility:

Unstable cardiac disease or any other medical condition likely to compromise the safe delivery of ChT or XRT; Clinically evident hearing impairment; Pre-existing motor or sensory neurotoxicity grade ≥ 2 according to the CTCAE v3.0;

* Any kind of previous therapy for SCCHN (excluding diagnostic biopsy)
* Previous administration of EGFR pathway-targeting therapy
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy which is not part of the study protocol
* Participation in another clinical trial within 30 days prior to study entry
* Pregnancy or breast feeding
* History of severe acute pulmonary disease
* Any investigational agent within past 30 days
* Other previous malignancy within 5 years, with exception of a history of a previously adequately treated basal cell carcinoma of the skin or pre- invasive carcinoma of the cervix
* Known drug abuse / severe alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent
* Active, uncontrolled infection
* Other medical condition or other therapy that in the opinion of the investigator precludes the safe administration of the planned ChT and XRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2011-10-30 (Actual)

PRIMARY OUTCOMES:
locoregional control | at 2 years post-therapy

SECONDARY OUTCOMES:
feasibility (toxicity profile) of the proposed regimen | during therapy
complete response rate | after induction ChT and 14-16 weeks after the therapy
disease free survival | at 2 years post-therapy
overall survival | at 2 years post-therapy
late toxicity including thyroid function | up to 2 years post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Primož Strojan, MD, Principal Investigator — Dept. of Radiation Oncology, Institute of Oncology Ljubljana, Slovenia
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia